CLINICAL TRIAL: NCT01112423
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Randomized, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of BMS-823778 in Non-Diabetic Subjects With Primary Hypercholesterolemia on a Stable Dose of Statin Therapy With or Without Ezetimibe
Brief Title: Safety Study of BMS-823778 in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB121-003
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — BMS-823778

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-823778 (2 mg) (Experimental)
  Interventions: Drug: BMS-823778
- BMS-823778 (10 mg) (Experimental)
  Interventions: Drug: BMS-823778
- BMS-823778 (20 mg) (Experimental)
  Interventions: Drug: BMS-823778
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-823778 — Capsules, Oral, 2 mg, once daily, 28 days
  Arms: BMS-823778 (2 mg)
Drug: BMS-823778 — Capsules, Oral, 10 mg, once daily, 28 days
  Arms: BMS-823778 (10 mg)
Drug: BMS-823778 — Capsules, Oral, 20 mg, once daily, 28 days
  Arms: BMS-823778 (20 mg)
Drug: Placebo — Capsules, Oral, 0 mg, once daily, 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacodynamic effects on LDL cholesterol (LDL-C)

ELIGIBILITY:
Inclusion Criteria:

* Hypercholesterolemia
* Currently taking a stable daily dose of statin therapy
* Serum triglyceride level < 500mg/dl

Exclusion Criteria:

* History of myocardial infarction, coronary angioplasty or bypass grafts, valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accidents within six months prior to entry into the study
* Congestive heart failure
* Diabetes mellitus
* Active liver disease
* Impaired renal function
* Hepatitis C, B and HIV

This list is not inclusive; additional information is provided in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Lowering of LDL-C | Within 28 days following dosing

SECONDARY OUTCOMES:
Pharmacokinetics (measuring trough concentrations) | On days 7, 14, and 28
Pharmacodynamic effects of BMS-823778 on Total cholesterol, HDL-C, Triglycerides, non-HDL-C, free fatty acids, Apolipoprotein fractions, HPA axis marker and free testosterone and sex hormone binding globulin (SHBG) | Within 28 days following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (6):
  - Osborne Research Center, Little Rock, Arkansas
  - Pra International, Lenexa, Kansas
  - Sterling Research Grp, Ltd., Cincinnati, Ohio
  - Cetero Research - San Antonio, San Antonio, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
- Local Institution, Brisbane, Queensland, Australia
- Canada (5):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, London, Ontario
  - Local Institution, Drummondville, Quebec
  - Local Institution, Montreal, Quebec

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx